CLINICAL TRIAL: NCT00077610
Title: A Randomized, Controlled, Open-label, Multi-center, Parallel-group Study to Demonstrate the Efficacy and Safety of RO0503821 When Administered Intravenously for the Maintenance Treatment of Anemia in Patients With Chronic Kidney Disease Who Are on Dialysis.
Brief Title: A Study of Intravenous Mircera for the Treatment of Anemia in Dialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA16739
Record Dates: First submitted 2004-02-10; First posted 2004-02-13 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-09

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa; Erythropoietin; continuous erythropoietin receptor activator

ARMS (3):
- RO0503821 (1x/2 Weeks) (Experimental): Participants received RO0503821 (Mircera [methoxy polyethylene glycol-epoetin beta]) once every two weeks intravenously for 52 weeks. Participants received a starting dose of RO0503821 (60, 100, or 180 microgram [mcg]) that was based on the Epoetin dose (<8000, 8000-16000, >16000 International units [IU]/Week) administered during the week preceding the switch to the study drug.
  Interventions: Drug: RO0503821 (1x/2 Weeks)
- RO0503821 (1x/4 Weeks) (Experimental): Participants received RO0503821 once every four weeks intravenously for 52 weeks. Participants received a starting dose of RO0503821 (120, 200, or 360 mcg) that was based on the Epoetin dose (<8000, 8000-16000, >16000 IU/Week) administered during the week preceding the switch to the study drug.
  Interventions: Drug: RO0503821 (1x/4 Weeks)
- Epoetin (1-3x/Weeks) (Active Comparator): Participants received their ongoing weekly intravenous dose of Epoetin alfa or beta one, two or three times weekly for 52 weeks.
  Interventions: Drug: Epoetin alfa or beta

INTERVENTIONS:
Drug: Epoetin alfa or beta — intravenously 3 times weekly for 52 weeks, as prescribed
  Other Names: Epoetin
  Arms: Epoetin (1-3x/Weeks)
Drug: RO0503821 (1x/2 Weeks) — 60, 100, or 180 microgram (mcg) (starting dose) once every two weeks intravenously for 52 weeks.
  Other Names: Mircera
  Arms: RO0503821 (1x/2 Weeks)
Drug: RO0503821 (1x/4 Weeks) — 120, 200 or 360 mcg (starting dose) once every four weeks intravenously for 52 weeks.
  Other Names: Mircera
  Arms: RO0503821 (1x/4 Weeks)

SUMMARY:
This study will assess the efficacy and safety of intravenous Mircera, given as maintenance treatment for renal anemia in chronic kidney disease patients on dialysis who were previously receiving iv epoetin. The anticipated time on study treatment is 1-2 years and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* chronic renal anemia;
* on dialysis therapy for at least 12 weeks before screening;
* receiving IV epoetin for at least 8 weeks before screening.

Exclusion Criteria:

* women who are pregnant, breastfeeding or using unreliable birth control methods;
* administration of another investigational drug within 4 weeks before screening, or during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 673 (Actual)
Dates: Start 2004-02; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (89):
- United States (54):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Montgomery, Alabama
  - Encino, California
  - Irvine, California
  - Los Angeles, California
  - Monterey Park, California
  - Riverside, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - San Jose, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Lakewood, Colorado
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Maywood, Illinois
  - Louisville, Kentucky
  - Covington, Louisiana
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Brooklyn Center, Minnesota
  - Paterson, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Great Neck, New York
  - Mineola, New York
  - New York, New York
  - Stony Brook, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Erie, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Orangeburg, South Carolina
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Burlington, Vermont
  - Fairfax, Virginia
  - Richmond, Virginia
  - Marshfield, Wisconsin
- Canada (8):
  - St. John's, Newfoundland and Labrador
  - Kingston, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Saskatoon, Saskatchewan
- France (5):
  - Aubervilliers
  - Bordeaux
  - La Tronche
  - Paris
  - Toulouse
- Germany (7):
  - Dortmund
  - Ellwangen
  - München
  - Nuremberg
  - Stuttgart
  - Wiesbaden
  - Wiesloch
- Italy (5):
  - Como
  - Lecco
  - Lodi
  - Milan
  - Pavia
- Norway (4):
  - Bergen
  - Levanger
  - Lillehammer
  - Trondheim
- Spain (5):
  - A Coruña
  - Barcelona
  - Madrid
  - Málaga
  - Seville
- Lausanne, Switzerland

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Levin NW, Fishbane S, Canedo FV, Zeig S, Nassar GM, Moran JE, Villa G, Beyer U, Oguey D; MAXIMA study investigators. Intravenous methoxy polyethylene glycol-epoetin beta for haemoglobin control in patients with chronic kidney disease who are on dialysis: a randomised non-inferiority trial (MAXIMA). Lancet. 2007 Oct 20;370(9596):1415-21. doi: 10.1016/S0140-6736(07)61599-2. PMID 17950856

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 673 participants were recruited at 91 centers in 8 countries with chronic renal anemia and dialysis therapy for at least 12 weeks before screening and during the screening/baseline period. This study was conducted between February 25, 2004 and August 17, 2005
Period: Overall Study
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin (1-3x/Weeks)
Started | 223 | 224 | 226
Started Treatment | 221 | 220 | 225
Completed | 169 | 168 | 180
Not Completed | 54 | 56 | 46
Not completed — Adverse Event | 9 | 7 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Withdrawal by Subject | 4 | 10 | 6
Not completed — Death | 17 | 13 | 13
Not completed — Renal transplant | 12 | 15 | 11
Not completed — Withdrew from dialysis care | 5 | 0 | 3
Not completed — Insufficient Therapeutic Response | 1 | 0 | 0
Not completed — Multiple blood transfusions | 0 | 0 | 1
Not completed — Principal Investigator's decision | 1 | 0 | 1
Not completed — Worsening of health condition | 1 | 1 | 0
Not completed — Given Epogen in hospital | 1 | 0 | 0
Not completed — Transferred to other unit | 0 | 0 | 1
Not completed — Transferred to nursing home | 0 | 0 | 1
Not completed — Transfer to satellite unit | 1 | 0 | 0
Not completed — Transfer to other center for surgery | 1 | 0 | 0
Not completed — Change in dialysis modality | 1 | 0 | 0
Not completed — Relocation | 0 | 8 | 5
Not completed — Financial issues | 0 | 1 | 0
Not completed — Sponsors decision to withdraw | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least one dose of RO0503821 or Epoetin, and a safety follow-up, whether withdrawn prematurely or not.
Groups:
- RO0503821 (1x/2 Weeks): Participants received RO0503821 once every two weeks intravenously for 52 weeks. Participants received a starting dose of RO0503821 (60, 100, or 180 mcg) that was based on the Epoetin dose (<8000, 8000-16000, >16000 IU/Week) administered during the week preceding the switch to the study drug.
- Total: Total of all reporting groups
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin (1-3x/Weeks) | Total
Number analyzed (Participants) | 221 | 220 | 225 | 666
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (15.05) | 59.0 (15.00) | 58.5 (15.16) | 58.9 (15.05)
Gender [Count of Participants; unit: Participants]
  Female | 89 | 95 | 92 | 276
  Male | 132 | 125 | 133 | 390

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin (Hb) Concentration From Baseline to Evaluation Period
Description: A time adjusted mean change in Hb concentration was calculated using an Area Under the Curve (AUC) approach, for both periods separately. Change in Hb concentration between the Baseline and evaluation periods was calculated by subtracting the calculated average baseline Hb from the average evaluation period Hb. At the end of the Week 36, data allowing the evaluation of the therapeutic response was available for 188 out of 221 eligible participants in RO0503821 (1x/2 Weeks) arm; 172 out of 220 eligible participants in RO0503821 (1x/4 Weeks); and 180 out of 225 participants in Epoetin (1-3x/Weeks) arm.
Time Frame: Baseline, Week 29 to Week 36
Population: The Per Protocol population included all randomized participants except those not meeting inclusion criterion related to Hb parameters and <5 recorded Hb values during the evaluation period with missing administrations of the study drug/ reference drug. Please refer to the outcome measure description section for more details.
Measure: Mean (Standard Deviation); unit: gram per deciliter (g/dL)
Groups:
- RO0503821 (1x/2 Weeks): Participants received RO0503821 once every two weeks intravenously for 52 weeks. Participants randomized received a starting dose of RO0503821 (60, 120,180 mcg) that was based on the Epoetin dose administered (<8000, 8000-16000, >16000 IU/Week) during the week preceding the switch to the study drug.
- RO0503821 (1x/4 Weeks): Participants received RO0503821 once every four weeks intravenously for 52 weeks. Participants randomized received a starting dose of RO0503821 (120, 200, 360 mcg) that was based on the Epoetin dose (<8000, 8000-16000, >16000 IU/Week) administered during the week preceding the switch to the study drug.
- Epoetin (1-3x/Week): Participants received their ongoing weekly intravenous dose of Epoetin alfa or beta one, two or three times weekly for 52 weeks.
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin (1-3x/Week)
Number analyzed (Participants) | 188 | 172 | 180
gram per deciliter (g/dL) | -0.10 (1.06) | 0.01 (0.96) | -0.10 (0.92)
Statistical Analysis 1: Comparison: RO0503821 (1x/2 Weeks) vs Epoetin (1-3x/Week); The non-inferiority test for treatment differences in Hb change from baseline, based on analysis of co-variance (ANCOVA) analysis with a non-inferiority limit of -0.75 g/dL; Test type: Non-Inferiority or Equivalence — The two RO0503821 dosing schedules were compared separately to epoetin reference using ANCOVA, with Hb at BL and region as the covariates. The test for non-inferiority was based on the lower limit of the two-sided 97.5% confidence interval for the difference between the two groups. When the lower limit was greater than or equal to -0.75 g/dL, the RO0503821 groups were regarded as non-inferior to the epoetin reference group. The confidence level of 97.5% was chosen to adjust for multiplicity; p < 0.0001, ANCOVA, CI for difference between groups; Mean Difference between groups = 0.004, 97.5% CI 2-sided [-0.215 to 0.223], Standard Error of Mean 0.0973 — Difference between groups based on the adjusted means derived from the ANCOVA model
Statistical Analysis 2: Comparison: RO0503821 (1x/4 Weeks) vs Epoetin (1-3x/Week); The non-inferiority test for treatment differences in Hb change from baseline, based on ANCOVA analysis with a non-inferiority limit of -0.75 g/dL; Test type: Non-Inferiority or Equivalence — The two RO0503821 dosing schedules were compared separately to epoetin reference using ANCOVA, with Hb at BL and region as the covariates. The test for non-inferiority was based on the lower limit of the two-sided 97.5% confidence interval for the difference between the two groups. When the lower limit was greater than or equal to -0.3 g/dL, the RO0503821 groups were regarded as non-inferior to the epoetin reference group. The confidence level of 97.5% was chosen to adjust for multiplicity; p < 0.0001, ANCOVA, CI for difference between groups; Mean Difference between groups = 0.051, 97.5% CI 2-sided [-0.173 to 0.275], Standard Error of Mean 0.0997 — Difference between groups based on the adjusted means derived from the ANCOVA model

2. Secondary Outcome: Number of Participants Maintaining Average Hemoglobin Concentration During Evaluation Period Within +/- 1 Gram Per Deciliter (g/dl) of Average Baseline Hemoglobin Concentration.
Description: The mean Hb of all values recorded during the evaluation period were calculated, and were subtracted from the mean baseline Hb for each participant. The number of participants maintaining their average Hb within +/- 1 g/dL of their average baseline hemoglobin concentration is given.
Time Frame: Baseline, Week 29 to Week 36
Population: The intent-to-treat (ITT) population was defined as all randomized participants. At the end of Week 36, data allowing the evaluation of the therapeutic response was available for 196/221, 188/220, and 205/225 participants in RO0503821 (1x/2 Weeks), RO0503821 (1x/4 Weeks), and Epoetin (1 -3x/Weeks), respectively.
Measure: Number; unit: participants
Groups:
- RO0503821 (1x/2 Weeks): Participants received RO0503821 once every two weeks intravenously for 52 weeks. Participants randomized received a starting dose of RO0503821 (60, 100,180 mcg) that was based on the Epoetin dose (<8000, 8000-16000, >16000 IU/Week) administered during the week preceding the switch to the study drug.
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin (1-3x/Weeks)
Number analyzed (Participants) | 196 | 188 | 205
participants | 133 | 127 | 138

3. Secondary Outcome: The Incidence of Red Blood Cell (RBC) Transfusions During the Titration and Evaluation Periods
Description: The number of participants who received RBC transfusions during the titration and evaluation periods were reported .
Time Frame: Week 1 to Week 36
Population: The Safety Population was defined as all participants who received at least one dose of RO0503821 or Epoetin, and a safety follow-up, whether withdrawn prematurely or not.
Measure: Number; unit: participants
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin (1-3x/Weeks)
Number analyzed (Participants) | 221 | 220 | 225
participants | 21 | 16 | 17

4. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in Platelet, White Blood Cell Counts (WBC) and Red Blood Cells (RBC)
Description: Marked laboratory abnormalities were defined as those values that were outside the Roche marked abnormality reference range. These abnormality laboratory values were flagged as Low or High if they were below the lower limit or above the upper limit of Roche marked abnormality reference range, respectively. The marked abnormality reference range for Platelet was 100-550x10^9/Litre [L], for WBC was 3.0-18.0.0x10^9/L, and for RBC was 3.80-6.10x10^12/L.
Time Frame: Up to Week 53
Population: The Safety Population was defined as all participants who received at least one dose of RO0503821 or Epoetin, and a safety follow-up, whether withdrawn prematurely or not. Participants available at particular time point were included in the analysis (n).
Measure: Number; unit: participants
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin (1-3x/Weeks)
Number analyzed (Participants) | 218 | 217 | 223
participants
  High Platelet (n=218, 216, 223) | 0 | 1 | 3
  Low Platelet (n=218, 216, 223) | 14 | 10 | 6
  High WBC (n=218, 217, 223) | 0 | 2 | 3
  Low WBC (n=218, 217, 223) | 8 | 6 | 5
  High RBC (n=124, 129, 89) | 1 | 2 | 0
  Low RBC (n=124, 129, 89) | 1 | 2 | 0

5. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities for Blood Chemistry and Electrolytes
Description: Marked laboratory abnormalities were defined as those values that were outside the Roche marked abnormality reference range. These abnormality laboratory values were flagged as Low or High if they were below the lower limit or above the upper limit of Roche marked abnormality reference range, respectively. The marked abnormality reference range for aspartate aminotransferase (AST) was 0-80 (unit per litre [U/L]), alanine aminotransferase (ALT) 0-110 U/L, alkaline phosphatase (ALP) 0-220 U/L, albumin >=30.0 gram/litre (g/L), glucose in non-diabetics 2.80-11.10 (millimol/litre [mmol/L]); potassium 2.90-5.80 mmol/L, and phosphorus 0.75-1.60 mmol/L
Time Frame: Up to Week 53
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin (1-3x/Weeks)
Number analyzed (Participants) | 218 | 216 | 224
participants
  High ALT. (n=218, 216, 224) | 4 | 2 | 5
  High ALP (n=218, 216, 224) | 15 | 14 | 16
  Low Albumin (n=218, 216, 224) | 14 | 13 | 18
  High Phosphate (n=218, 216, 224) | 106 | 95 | 94
  Low Phosphate (n=218, 216, 224) | 21 | 21 | 17
  High Potassium (n=218, 216, 224) | 33 | 35 | 36
  Low Potassium (n=218, 216, 224) | 10 | 3 | 3
  High AST (n=218, 215, 224) | 6 | 3 | 4
  High Blood glucose in non-diabetic (n=114,131,110) | 0 | 3 | 1
  Low Blood Glucose in Non-Diabetic (n=114,131,110) | 0 | 1 | 0

6. Secondary Outcome: Mean Change in Blood Pressure From Baseline at Week 36 and Week 52
Description: Blood pressure was measured by manual assessment or automated reading throughout the entire study for every participant. Blood pressure was taken in the sitting position after at least 5 minutes rest. An appropriate -sized cuff was used and both systolic (SBP) and diastolic (DBP) blood pressures were recorded before dialysis (BD) and after dialysis (AD).
Time Frame: Baseline, Week 36 and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin (1-3x/Weeks)
Number analyzed (Participants) | 189 | 178 | 196
millimeter of mercury (mmHg)
  Change in SBP, BD at Wk 36 (n=189, 178,196) | 1 (25.3) | -2 (22.7) | 3 (25.1)
  Change in SBP, BD at Wk 52 (n=168, 166, 180) | -0 (24.6) | -3 (24.6) | 1 (26.0)
  Change in DBP, BD at Wk 36 (n=189, 178, 195) | 0 (14.7) | -3 (16.3) | 1 (16.8)
  Change in DBP, BD at Wk 52 (n=168, 166, 179) | 1 (15.2) | -3 (18.3) | -1 (15.4)
  Change in SBP, AD at Wk 36 (n=189, 177, 196) | 3 (28.3) | -1 (27.0) | -0 (24.3)
  Change in SBP, AD at Wk 52 (n=167, 168, 179) | 2 (24.5) | -0 (29.3) | 1 (24.9)
  Change in DBP, AD at Wk 36 (n=189, 177, 196) | -1 (16.4) | -0 (15.2) | -2 (12.4)
  Change in DBP, AD at Wk 52 (n=167, 168, 178) | -1 (14.9) | -0 (15.9) | -3 (14.9)

7. Secondary Outcome: Mean Change in Pulse Rate (Sitting) From Baseline at Week 36 and Week 52
Description: Change in pulse rate (beats per minute [bpm]) from baseline values includes only those participants with both a baseline value and a value for specified time period.
Time Frame: Baseline, Week 36 and Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin (1-3x/Weeks)
Number analyzed (Participants) | 188 | 176 | 193
beats per minute (bpm)
  Change from BL at Week 36 (n=188, 176, 193) | 1 (12.0) | 2 (11.8) | 0 (14.5)
  Change from BL at Week 52 (n=168, 166, 179) | 1 (13.6) | 1 (13.4) | -1 (13.2)

8. Secondary Outcome: Incidence of Adverse Events (AEs), Serious Adverse Events (SAEs) and Death
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is a significant medical event in the investigator's judgment or requires intervention to prevent one or other of these outcomes. Overall deaths occurred in the study were reported.
Time Frame: Upto Week 53
Population: as for outcome 4
Measure: Number; unit: participants
Groups:
- RO0503821 (1x/4 Weeks): Participants received RO0503821 once every four weeks intravenously for 52 weeks. Participants randomized received a starting dose of RO0503821 (120, 200, 360 mcg) that was based on the Epoetin dose administered during the week preceding the switch to the study drug.
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin (1-3x/Weeks)
Number analyzed (Participants) | 221 | 220 | 225
participants
  Number of participants with adverse events | 203 | 202 | 214
  Number of participants with serious adverse events | 101 | 87 | 99
  Number of deaths | 19 | 15 | 17

ADVERSE EVENTS:
Time Frame: Up to Week 53
Description: Of 673 recruited participants, 7 withdrew before receiving the study drug (2 in the RO0503821 [1x/2 Weeks], 4 in the RO0503821 [1x/4 Weeks] and 1 from Epoetin group). The safety population included all participants who received at least one dose of RO0503821 or Epoetin, and a safety follow-up, whether withdrawn prematurely or not.
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin (1-3x/Weeks)
Serious Adverse Events (participants affected / at risk) | 101/221 | 87/220 | 99/225
Other Adverse Events (participants affected / at risk) | 166/221 | 151/220 | 175/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (1x/2 Weeks) (N=221) | RO0503821 (1x/4 Weeks) (N=220) | Epoetin (1-3x/Weeks) (N=225)
Sepsis (Infections and infestations) | 5 | 6 | 9
Pneumonia (Infections and infestations) | 9 | 5 | 5
Cellulitis (Infections and infestations) | 3 | 1 | 4
Arteriovenous graft site infection (Infections and infestations) | 1 | 3 | 2
Staphylococcal bacteraemia (Infections and infestations) | 2 | 3 | 1
Gangrene (Infections and infestations) | 1 | 0 | 3
Septic shock (Infections and infestations) | 0 | 2 | 2
Staphylococcal sepsis (Infections and infestations) | 2 | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 2
Urosepsis (Infections and infestations) | 0 | 3 | 0
Catheter sepsis (Infections and infestations) | 1 | 1 | 0
Clostridium colitis (Infections and infestations) | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1
Lobar pneumonia (Infections and infestations) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Arteriovenous graft site abscess (Infections and infestations) | 1 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Bronchitis acute viral (Infections and infestations) | 0 | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0
Postoperative infection (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Sepsis syndrome (Infections and infestations) | 0 | 0 | 1
Splenic abscess (Infections and infestations) | 0 | 1 | 0
Staphylococcal osteomyelitis (Infections and infestations) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 6 | 3 | 7
Myocardial infarction (Cardiac disorders) | 3 | 3 | 7
Cardiac arrest (Cardiac disorders) | 8 | 2 | 2
Cardio respiratory arrest (Cardiac disorders) | 3 | 2 | 3
Acute myocardial infarction (Cardiac disorders) | 3 | 2 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 4 | 1
Coronary artery disease (Cardiac disorders) | 3 | 0 | 3
Aortic valve stenosis (Cardiac disorders) | 1 | 3 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 2
Angina unstable (Cardiac disorders) | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Aortic valve calcification (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 2 | 8 | 7
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 | 4 | 4
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 2 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 2 | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal dilatation (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal infarction (Endocrine disorders) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 5 | 4 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 2
Hypertensive crisis (Vascular disorders) | 1 | 1 | 2
Peripheral ischaemia (Vascular disorders) | 0 | 3 | 1
Hypertension (Vascular disorders) | 1 | 1 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0
Venous stenosis (Vascular disorders) | 1 | 0 | 1
Air embolism (Vascular disorders) | 1 | 0 | 0
Aneurysm arteriovenous (Vascular disorders) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 0 | 1
Arteriovenous fistula (Vascular disorders) | 0 | 1 | 0
Diabetic vascular disorder (Vascular disorders) | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 0 | 0
Haematoma (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Hypoperfusion (Vascular disorders) | 0 | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
Vascular pseudoaneurysm (Vascular disorders) | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0
Wound haemorrhage (Vascular disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 2 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 1 | 1
Cerebral thrombosis (Nervous system disorders) | 0 | 3 | 0
Dementia (Nervous system disorders) | 1 | 0 | 1
Benign intracranial hypertension (Nervous system disorders) | 0 | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Complex partial seizures (Nervous system disorders) | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Syncope vasovagal (Nervous system disorders) | 1 | 0 | 0
Thrombotic stroke (Nervous system disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 2 | 7
Non-cardiac chest pain (General disorders) | 2 | 1 | 2
Multi-organ failure (General disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 1 | 0
Sudden death (General disorders) | 0 | 2 | 0
Catheter related complication (General disorders) | 0 | 0 | 1
Catheter site haemorrhage (General disorders) | 1 | 0 | 0
Hyperpyrexia (General disorders) | 0 | 1 | 0
Hypothermia (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Intervertebral discitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bursa disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 4 | 1 | 7
Haematuria (Renal and urinary disorders) | 2 | 0 | 0
Renal disorder (Renal and urinary disorders) | 1 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 2 | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 1 | 1
Hypomania (Psychiatric disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Diabetic dermopathy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 1 | 0
Kidney transplant rejection (Immune system disorders) | 0 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Angle closure glaucoma (Eye disorders) | 0 | 0 | 1
Blindness transient (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1
Female genital-digestive tract fistula (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 1 | 0
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0
Vestibular neuronitis (Ear and labyrinth disorders) | 1 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0
Renal haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (1x/2 Weeks) (N=221) | RO0503821 (1x/4 Weeks) (N=220) | Epoetin (1-3x/Weeks) (N=225)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 24 | 23 | 28
Fall (Injury, poisoning and procedural complications) | 15 | 19 | 15
Procedural hypotension (Injury, poisoning and procedural complications) | 18 | 20 | 9
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 16 | 10 | 15
Vascular graft complication (Injury, poisoning and procedural complications) | 8 | 13 | 13
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 9 | 8 | 15
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 12 | 7 | 4
Nasopharyngitis (Infections and infestations) | 28 | 39 | 24
Upper respiratory tract infection (Infections and infestations) | 20 | 30 | 25
Urinary tract infection (Infections and infestations) | 13 | 12 | 9
Gastroenteritis (Infections and infestations) | 6 | 11 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 | 19 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 11 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 15 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 3 | 12
Diarrhoea (Gastrointestinal disorders) | 37 | 25 | 30
Vomiting (Gastrointestinal disorders) | 16 | 11 | 14
Nausea (Gastrointestinal disorders) | 10 | 9 | 15
Constipation (Gastrointestinal disorders) | 12 | 4 | 12
Headache (Nervous system disorders) | 30 | 17 | 24
Dizziness (Nervous system disorders) | 6 | 13 | 12
Pyrexia (General disorders) | 8 | 8 | 17
Asthenia (General disorders) | 11 | 15 | 6
Fatigue (General disorders) | 12 | 9 | 6
Hypertension (Vascular disorders) | 22 | 28 | 34
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 19 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 15
Fluid overload (Metabolism and nutrition disorders) | 23 | 18 | 13
Insomnia (Psychiatric disorders) | 11 | 14 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 11 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.